CLINICAL TRIAL: NCT03083951
Title: Complete Mesocolon Excision vs Locoregional Lymphadenectomy in Sigmoid Colon Cancer (CMELL)
Acronym: CMELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pere Planellas Giné (Other)
Responsible Party: Sponsor-Investigator, Pere Planellas Giné, Principal investigator, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Organization: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13117
Record Dates: First submitted 2017-03-02; First posted 2017-03-20 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer; Sigmoid Cancer
Keywords: Complete mesocolon excision; Sigmoid cancer; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Sigmoid Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, single blind (the patient does not know the group to which it has been assigned) of patients undergoing laparoscopic sigmoid colon cancer resection. In all patients a lymphadenectomy with a high ligation of the Lower Mesenteric Artery will be performed. In patients in group 1A, lymphadenectomy will also include the lymphogranular tissue that accompanies the inferior mesenteric vein from its origin (complete mesocolon excision). In patients in group 1B, a conventional lymphadenectomy will be performed only from the origin of the inferior mesenteric artery without including the lymphatic tissue of the origin of the inferior mesenteric vein.
Who Masked: Participant
Masking Description: The patient does not know the group to which it has been assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complete Mesocolon Excision (Experimental): A high tie of the inferior mesenteric artery (IMA) should be attempted. The inferior mesenteric vein section at the Treitz angle should be performed. The lymphatic tissue that accompanies the inferior mesenteric vein should be added.
  Interventions: Procedure: Complete mesocolon excision
- Conventional Locoregional Lymphadenectomy (Active Comparator): A high tie of the inferior mesenteric artery (IMA) should be attempted. Lymphadenectomy of the lymphatic tissue that accompanies the IMA will be performed. The inferior mesenteric vein section could be performed at the discretion of the surgeon.
  Interventions: Procedure: Conventional locoregional lymphadenectomy

INTERVENTIONS:
Procedure: Complete mesocolon excision — Laparoscopic sigmoidectomy with lymphadenectomy of the lymphatic tissue that accompanies the inferior mesenteric vein and a high tie ligation of the inferior mesenteric artery (complete mesocolon excision)
  Arms: Complete Mesocolon Excision
Procedure: Conventional locoregional lymphadenectomy — Laparoscopic sigmoidectomy with lymphadenectomy of the lymphatic tissue that accompanies the inferior mesenteric artery and a high tie ligation of the inferior mesenteric artery with or without section of inferior mesenteric vein.
  Arms: Conventional Locoregional Lymphadenectomy

SUMMARY:
A randomized, controlled clinical trial comparing lymphadenectomy with extended inferior mesenteric artery ligation (complete mesocolon excision: which includes lymphoma tissue from the origin of the inferior mesenteric vein) with conventional locoregional lymphadenectomy in patients undergoing laparoscopic sigmoidectomy for sigmoid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing programmed surgery for laparoscopic sigmoid colon cancer.
* Age ≥ 18 years and <80 years.
* Histology of adenocarcinoma or adenoma without chemotherapy or neoadjuvant radiotherapy.
* Any T, any N, M0.
* Intention of resection R0.
* Informed consent signed by the patient and the investigator.

Exclusion Criteria:

* Colorectal tumor with histology other than adenocarcinoma or adenoma.
* Colon cancer located in the right colon, transverse, splenic or non-sigmoid left colon.
* Metastatic disease (M1).
* History of colorectal cancer surgery, different from a local excision.
* Inflammatory bowel disease with anatomopathological confirmation.
* Patients with psychiatric illness, addiction or any disorder that impedes the understanding of informed consent.
* Inability to read or understand any of the languages of the informed consent (Catalan, Spanish).
* Another synchronous malignant disease.
* Emergency surgery.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Total number of lymph nodes and lymph node ratio. | 30 days
  To compare the total number of lymph nodes resected and the lymph node ratio (defined as ratio of lymph nodes with tumor metastasis to the total lymph nodes resected) between the two arms.

SECONDARY OUTCOMES:
Local recurrence | 5 years
  To compare the tumor local recurrence rate between the two arms.
Survival | 5 years
  To compare the survival rate (deaths from cancer) between the two arms

OTHER OUTCOMES:
Postoperative complications | 90 days
  Postoperative complications within 90 days after surgery (Clavien-Dindo classification).
Anastomotic leakage | 90 days
  To compare the incidence of anastomotic leakage according to the classification of the International Group for Rectal Cancer Study.
Intraoperative outcomes: duration of surgery | 1 day
  To compare the duration of surgery measured in minutes between the two arms
Intraoperative outcomes: surgical bleeding | 1 day
  To compare the surgical bleeding measured in ml between the two arms
Intraoperative outcomes: surgical conversion | 1 day
  To compare the incidence of surgical conversion to laparotomy between the two arms
Genitourinary dysfunction assessed by ICIQ-SF questionnaire | 1 year
  To compare the Genitourinary dysfunction between the two arm measured by ICIQ-SF questionnaire
Defecatory dysfunction assessed by FSFI and erectile dysfunction questionnaires | 1 year
  To compare the defecatory dysfunction between the two arms measured by FSFI and erectile dysfunction questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Dr. Josep Trueta of Girona, Girona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Planellas P, Marinello F, Elorza G, Golda T, Farres R, Espin-Basany E, Enriquez-Navascues JM, Kreisler E, Cornejo L, Codina-Cazador A. Impact on defecatory, urinary and sexual function after high-tie sigmoidectomy: a post-hoc analysis of a multicenter randomized controlled trial comparing extended versus standard complete mesocolon excision. Langenbecks Arch Surg. 2023 Aug 1;408(1):293. doi: 10.1007/s00423-023-03026-9. PMID 37526748
- [Derived] Planellas P, Marinello F, Elorza G, Golda T, Farres R, Espin-Basany E, Enriquez-Navascues JM, Kreisler E, Cornejo L, Codina-Cazador A. Extended Versus Standard Complete Mesocolon Excision in Sigmoid Colon Cancer: A Multicenter Randomized Controlled Trial. Ann Surg. 2022 Feb 1;275(2):271-280. doi: 10.1097/SLA.0000000000005161. PMID 34417367